CLINICAL TRIAL: NCT00859742
Title: Endobronchial Ultrasound Guided Transbronchial Needle Aspiration for the Mediastinal Re-staging After Induction Therapy in Non-small Cell Lung Cancer. A Prospective Study
Brief Title: Endobronchial Ultrasound Guided Transbronchial Needle Aspiration (EBUS-TBNA) for Mediastinal Re-staging of Non-small Cell Lung Cancer(NSCLC)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Bin Hwangbo, Principal Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCCTS-06-211
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EBUS-TBNA (Experimental)
  Interventions: Procedure: EBUS-TBNA, integrated PET/CT

INTERVENTIONS:
Procedure: EBUS-TBNA, integrated PET/CT — EBUS-TBNA and integrated PET/CT will be performed for patients with non-small cell lung cancer after induction therapy. PET/CT will be performed before EBUS-TBNA. Negative findings of EBUS-TBNA will be evaluated by surgery.

SUMMARY:
The aim of this study is to determine the diagnostic values of EBUS-TBNA in the mediastinal re-staging after induction treatment in patients with non-small cell lung cancer.

Primary objective:

1. To determine the sensitivity, specificity, positive predictive value, negative predictive value and the accuracy of EBUS-TBNA in the detection of mediastinal metastasis in mediastinal re-staging after induction treatment.

Secondary objectives:

1. To compare the diagnostic values of EBUS-TBNA and integrated PET/CT in mediastinal re-staging
2. To evaluate the changes of ultrasonographic features of mediastinal lymph nodes after induction therapy
3. To determine procedure related complications

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-small cell lung cancer
* Patients who have initially histologically proven N2 disease (Stage IIIA)
* Patients who underwent induction treatment (chemotherapy or chemoradiation therapy) and are considred for surgery
* Written informed consent

Exclusion Criteria:

* Contraindications for bronchoscopy
* Medically inoperable patients
* Patients who are found to have M1 disease, inoperable T4 disease or supraclavicular metastasis after induction treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
The diagnostic values of EBUS-TBNA in the mediastinal re-staging after induction treatment in non-small cell lung cancer. | 1.5 years

SECONDARY OUTCOMES:
The diagnostic values of integrated PET/CT in the mediastinal re-staging after induction treatment in non-small cell lung cancer | 1.5 years
The changes of ultrasonographic features of mediastinal lymph nodes after induction therapy | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bin Hwangbo, MD. PhD, Principal Investigator — Goyang, Gyeonggi-do, Korea, Republic of
Locations (1):
- NCCKorea, Goyang-si, Gyeonggi-do, South Korea